CLINICAL TRIAL: NCT04523818
Title: A Phase Ib Trial of Preoperative Short-Course Chemoradiotherapy Followed by Chemotherapy for Resectable Gastric Adenocarcinoma
Brief Title: Short-Course Chemoradiotherapy Followed by Chemotherapy for the Treatment of Resectable Gastric Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0481; NCI-2020-05810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0481 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Gastric Adenocarcinoma; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage I Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage II Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage III Gastric Cancer AJCC v8
MeSH Terms: interventions — Capecitabine; Fluorouracil; dehydroftorafur; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CXRT, chemotherapy, surgery) (Experimental): Patients receive CXRT consisting of radiation therapy 5 days a week (Monday through Friday) for 2 weeks (10 treatments) and standard of care chemotherapy consisting of capecitabine PO BID or fluorouracil IV continuous Monday to Friday of each radiation week. About 2 weeks later, patients receive standard of care chemotherapy for up to 2 months in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery 3-8 weeks post-chemotherapy completion.
  Interventions: Drug: Capecitabine; Drug: Fluorouracil; Radiation: Radiation Therapy; Procedure: Therapeutic Surgical Procedure

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Surgical Procedure — Undergo standard of care surgery

SUMMARY:
This phase Ib trial investigates the side effects and how well a shorter course of chemotherapy and radiation treatment (chemoradiotherapy) for 2 weeks instead of 5 weeks followed by standard chemotherapy works in treating patients with gastric cancer who are scheduled to have treatment and then surgery to remove the tumor. Chemotherapy drugs, such as capecitabine and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy sources to kill tumor cells and shrink tumors. Giving short-course chemo-radiotherapy before chemotherapy and surgery may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of preoperative short-course chemoradiotherapy (CXRT) in patients with potentially resectable gastric adenocarcinoma.

SECONDARY OBJECTIVES:

I. To assess the rate of pathologic complete response (pathCR) in patients treated with preoperative short-course CXRT.

II. To assess the rate of perioperative complications after gastrectomy in patients treated with preoperative short-course CXRT.

III. To assess overall survival from the date of diagnosis in subjects treated with short course CXRT.

OUTLINE:

Patients receive CXRT consisting of radiation therapy 5 days a week (Monday through Friday) for 2 weeks (10 treatments) and standard of care chemotherapy consisting of capecitabine orally (PO) twice daily (BID) or fluorouracil intravenously (IV) continuous Monday to Friday of each radiation week. About 2 weeks later, patients receive standard of care chemotherapy for up to 2 months in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery 3-8 weeks post-chemotherapy completion.

After the completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients with a biopsy-confirmed diagnosis of adenocarcinoma of the stomach
* No evidence of distant metastatic disease based on standard of care preoperative imaging evaluation
* Evidence of T2 stage or greater primary tumor, or any T stage with node positive disease based on endoscopic ultrasound or standard of care imaging
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,500/ul
* Platelets >= 60,000/UI
* Glomerular filtration rate >= 60 mL/min/1.73 m^2. The estimated glomerular filtration rate (eGFR) is calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. The eGFR declines with age. eGFR < 60 mL/min/1.73 m2 is considered as "decreased". This equation should only be used for patients 18 and older. According to the National Kidney Foundation's Kidney Disease Outcome Quality Initiative (KDOQI) classification and 2012 Kidney Disease Improving Global Outcomes (KDIGO) Clinical Practice Guideline, the stage of CKD should be categorized based on estimated GFR

Exclusion Criteria:

* Presence of metastatic disease on staging with standard of care imaging, with or without diagnostic laparoscopy. Subjects not able to undergo staging laparoscopy due to previous surgery will not be excluded from this trial, and the determination of absence of metastatic disease will be decided solely on imaging consistent with our current standard of care
* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract
* Infections such as pneumonia or wound infections that would preclude protocol therapy
* Women with a positive urine or serum pregnancy test are excluded from this study; women of childbearing potential (defined as those who have not undergone a hysterectomy or who have not been postmenopausal for at least 12 consecutive months) must agree to refrain from breast-feeding and practice adequate contraception as specified in the informed consent. Adequate contraception consists of oral contraceptive, implantable contraceptives, injectable contraceptives, barrier methods, or abstinence. Contraception for males consists of barrier methods or abstinence
* Subjects with unstable angina or New York Heart Association grade II or greater congestive heart failure
* Subjects deemed unable to comply with study and/or follow-up procedures
* Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity
* Prior radiotherapy to the same field
* Comorbid conditions (examples - collagen vascular diseases, certain genetic conditions that predispose to secondary malignancies) that are prohibitive to preoperative therapy, or contraindications to radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 4 weeks following last chemotherapy
  Characterized by the incidence and severity of treatment-related adverse events. Grade 3 or higher toxicity classified as attributable to chemotherapy and radiation treatment (CXRT), during the 14 days of treatment administration or within 14 days of completion of CXRT (i.e., a total of 28 days), based on multidisciplinary review, will be used for the purpose of toxicity monitoring. Differences between grades vary and are detailed according to the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. In general, Grade 3 toxicity refers to any event that requires hospitalization with intervention (i.e., intravenous [IV] hydration, symptomatic control, transfusion, procedure, etc.).

SECONDARY OUTCOMES:
Rate of pathologic complete response in patients treated with resection | Up to 5 years
  Will be estimated, along with exact 95% confidence intervals.
Rate of perioperative complications after gastrectomy in patients treated with preoperative short course CXRT and chemotherapy | Up to 5 years
  Will be estimated, along with exact 95% confidence intervals.
Overall survival (OS) | Up to 5 years
  Will be evaluated using the Kaplan-Meier method. Median OS and the 95% confidence interval will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Badgwell, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT04523818/ICF_000.pdf